CLINICAL TRIAL: NCT03163251
Title: The Reflect, Empathize, Analyze, and Discuss in Small Groups Study: The Effect of Peer-facilitated Small Group Discussions on Burnout and Professional Development Among Physician Trainees
Brief Title: The READ-SG Study: Effect of Peer-Facilitated Small Group Discussions
Acronym: READ-SG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAP0006
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Burnout, Professional; Emotional Intelligence; Peer Influence
Keywords: READ-SG; Burnout; Professional identity; Empathy; Emotional intelligence
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: This is a single institution, single arm, prospective cohort study stratified by post-graduate training year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- READ-SG Cohort (Experimental): Each post-graduate year (PGY) will receive the intervention of a monthly peer-facilitated small group sessions (READ-SG Sessions) based on topics that are common to residency training and based on themes regarding humanism in medicine.
  Interventions: Behavioral: READ-SG Sessions

INTERVENTIONS:
Behavioral: READ-SG Sessions — In the Internal Medicine residency program at Columbia University Medical Center, PGY-1 trainees receive an hour of protected time to attend a monthly peer-facilitated small group session, outlined above. PGY-2 and 3 trainees have a similar combined session separate from the PGY-1s. Facilitators are chosen by the READ-SG Committee, which is comprised of Mark P. Abrams (Director, Co-Investigator), Evelyn Granieri (Faculty Advisor, PI), a Chief Resident from the program (Program Liaison), and the facilitators.
  Other Names: READ-SG

SUMMARY:
This study evaluates the effect of peer facilitated monthly small group topic-based small group discussions on various themes common to physician training that pertain to aspects of humanism on rates of burnout. Attendance to these sessions and completion of the surveys is voluntary.

DETAILED DESCRIPTION:
It is widely known that physicians have rates of suicide that are far higher than in other professions: 70% higher for men and 250-400% higher for women. While the reasoning behind why this occurs has not been well elucidated, physicians do face some unique challenges including the responsibilities of the lives of others, a duty to always uphold the highest level of a moral and ethical standard, as well as being faced with both physical and emotional exhaustion. Trainees in particular seem at risk due to the rigors of the job in addition to the stress of the rapid expansion of the physical and emotional expectations put upon them.

To the investigator's knowledge, there has yet to be any study that has shown any beneficial outcomes regarding burnout using a small group curriculum among physician trainees that also encompasses analysis of the effect of an intervention on the emotional development of trainees. However, there has been a randomized trial on the effect of small groups for junior attendings that showed decreased rates of depersonalization, emotional exhaustion, and physician burnout in the intervention group. The implications of such programs on the trainee population could result in decreased levels of physician/ trainee burnout, depression, and potentially even suicide, aside from providing trainees with a sense of increased job satisfaction.

While many people in the scientific community judge the success of a physician by their medical achievements and diagnostic acumen, many patients judge the successes of their doctors based on empathy, communication, and bedside manner. While many resources exist to teach residents about the science of medicine, there does not exist to my knowledge a standardized curriculum to teach residents about the humanistic side of medicine and the importance of emotional development. Implementing such a curriculum could provide exactly what is missing from formal residency training as it stands now. Such a program that could be easily adapted to a large number of trainees would seem to be beneficial and also be in line with the Accreditation Council for Graduate Medical Education (ACGME)'s core competencies intended for residents to improve on patient care, professionalism, and interpersonal communication.

Peer support and teamwork seem like logical coping mechanisms for a vulnerable population that can feel isolated, such as physician trainees. The study aims to elucidate whether the peer-facilitated READ-SG method is effective at reducing burnout, as assessed by the Maslach Burnout Inventory, the gold standard in the field of assessing burnout, as well as to gauge the perceived effect of each session on participants' professional development and symptoms of burnout.

ELIGIBILITY:
Inclusion Criteria:

- Internal Medicine trainees in the PGY-1 through PGY-3 years at New York Presbyterian - Columbia University Medical Center.

Exclusion Criteria:

- Not open to anyone outside of the Internal Medicine trainees at New York Presbyterian - Columbia University Medical Center.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Maslach Burnout Inventory-Human Services Survey (MBI-HSS) Personal Accomplishment Score (section 1) | Baseline, 1 year
  This is designed to prospectively measure whether the intervention affects and/or mitigates burnout rates over residency training. The survey has 3 sections.
Change in Maslach Burnout Inventory-Human Services Survey (MBI-HSS) Depersonalization Score (section 2) | Baseline, 1 year
  This is designed to prospectively measure whether the intervention affects and/or mitigates burnout rates over residency training. The survey has 3 sections.
Change in Maslach Burnout Inventory-Human Services Survey (MBI-HSS) Emotional Exhaustion Score (section 3) | Baseline, 1 year
  This is designed to prospectively measure whether the intervention affects and/or mitigates burnout rates over residency training. The survey has 3 sections.

SECONDARY OUTCOMES:
Dose response relationship ratio | Up to 1 year
  This is designed to evaluate whether there is a dose response relationship between the number of sessions attended and the effect of the sessions on burnout scores, measured by p-value.
Change in Likert-scale Score | Baseline, monthly for up to 1 year
  This is designed to validate whether the READ-SG Study Survey correlate with the already validated single-question/abbreviated burnout questions.

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Abrams, MD, Study Director — Postdoctoral Clinical Fellow in the Department of Medicine, Dept of Medicine Cardiology; Evelyn Granieri, MD, Principal Investigator — Professor of Medicine at the Columbia University Medical Center, Dept of Medicine Geriatrics
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] West CP, Dyrbye LN, Rabatin JT, Call TG, Davidson JH, Multari A, Romanski SA, Hellyer JM, Sloan JA, Shanafelt TD. Intervention to promote physician well-being, job satisfaction, and professionalism: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):527-33. doi: 10.1001/jamainternmed.2013.14387. PMID 24515493
- [Background] Abrams MP, Granieri E. Peer facilitation and burnout: the READ-SG pilot. Clin Teach. 2018 Jun;15(3):226-230. doi: 10.1111/tct.12666. Epub 2017 May 10. PMID 28493398
- [Background] Abrams MP. Improving Resident Well-Being and Burnout: The Role of Peer Support. J Grad Med Educ. 2017 Apr;9(2):264. doi: 10.4300/JGME-D-16-00805.1. No abstract available. PMID 28439373